CLINICAL TRIAL: NCT01022268
Title: A Comprehensive, Long-term Integrated Programme to Study the Aetiology and Immunopathology of Childhood Infectious, Inflammatory and Allergic Disease, Using the Large Patient Base of Children Attending St Mary's Hospital, London
Brief Title: Understanding Childhood Infection, Inflammation and Allergy
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1330
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-04

CONDITIONS: Infection; Inflammation; Allergy; Children
Keywords: Inflammation; Children; Observational
MeSH Terms: conditions — Infections; Inflammation; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma DNA RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection, inflammation or allergy: Children presenting via any means to St Mary's Hospital; this would include the A&E department, the general and infectious disease wards and the paediatric intensive care unit.
  Children needing blood tests for any clinical reason Children who, in the clinical judgement of the doctor assessing them, have presented because of a condition consistent with an infectious, inflammatory or allergic process
- controls: children who do not have an infectious, inflammatory or allergic condition, who anyway require blood tests for clinical reasons

SUMMARY:
This proposal represents a unified programme supported by both clinical and academic staff in the Departments of Paediatrics at Imperial College and St Mary's Hospital, Southampton Hospital and John Radcliffe Hospital (Oxford). St Mary's Hospital is the hub of a paediatric network for West London, and forms part of the Paediatric Intensive Care Network for the London region, with potential access to a population of 3 million children.

We aim to improve diagnosis and understanding of children with infectious, inflammatory and allergic conditions. Our study will establish well-characterised cohorts of patients with defined conditions, in whom microbiological and patient samples will be used to understand the contribution of genetic background, differential gene expression, proteomics and the pathogen type to the disease process.

Unwell children coming to hospital through any route will be invited to join the study. Entering the study will entail the child having blood taken for research purposes in addition to the clinically indicated tests. We will also recruit well (control) children who are having blood tests performed for elective purposes, such as surgery.

In addition, children presenting with an illness that is likely to have an infectious aetiology will also have samples collected for microbiological diagnosis. Those samples taken for ordinary diagnostic purposes (such as blood, urine, cerebrospinal fluid (CSF), bronchoalveolar lavage (BAL) fluid or nasal brushings for epithelial cell cultures) would also be used for state-of-the-art diagnostic techniques, in order to maximise the likelihood of confirming a microbiological diagnosis. Where healthy, uninfected children are having invasive procedures, such as lumbar punctures, we would aim to recruit these children as controls and collect biological samples such as CSF samples.

This bid addresses the need for translational research in paediatrics, by building on the world-class basic science and clinical paediatric base at Imperial College and St Mary's Hospital.

DETAILED DESCRIPTION:
There is currently little understanding of the mechanisms by which respiratory infections can cause severe illness and death. The emergence of Influenza A subtype (H1N1) as a major cause of childhood severe illness in 2009 permitted further study of how this virus triggers severe disease, and how the inflammatory response to H1N1 differs from other infections. It is likely that host-mediated inflammatory processes triggered by the infecting agent contributes to severe illness. In addition, viral infection induces profound changes in the innate immune response to common bacterial pathogens, with increased bacterial colonisation of normally sterile lower airway. Thus both host and bacterial factors may contribute to lung damage in severe respiratory infection.

This study was initiated to identify the aetiology and immunopathologic mechanisms of childhood respiratory infection (Immunopathology of Respiratory Infection Study - IRIS), recruiting children with suspected respiratory infection or respiratory failure (and controls). This dataset will provide a unique resource for further study of disease mechanisms in children with a range of infections including H1N1/09 infection, Respiratory Syncytial Virus (RSV), Rhinovirus, other common respiratory viruses and severe bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* children presenting via any means to Hospital
* children needing blood tests for any clinical reason
* children who have presented because of a condition consistent with an infectious, inflammatory or allergic process

Exclusion Criteria:

* aged 17 or older
* children re-presenting with the same condition
* concern that the study is not fully understood by the parent or guardian

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Unwell children coming to St Mary's Hospital, Southampton Hospital or John Radcliffe Hospital (Oxford) through any route (Emergency Department, wards, intensive care)
Sampling Method: Non-Probability Sample
Enrollment: 902 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, Paddington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cebey-Lopez M, Herberg J, Pardo-Seco J, Gomez-Carballa A, Martinon-Torres N, Salas A, Martinon-Sanchez JM, Gormley S, Sumner E, Fink C, Martinon-Torres F; GENDRES network. Viral Co-Infections in Pediatric Patients Hospitalized with Lower Tract Acute Respiratory Infections. PLoS One. 2015 Sep 2;10(9):e0136526. doi: 10.1371/journal.pone.0136526. eCollection 2015. PMID 26332375
- [Background] Cebey-Lopez M, Herberg J, Pardo-Seco J, Gomez-Carballa A, Martinon-Torres N, Salas A, Martinon-Sanchez JM, Justicia A, Rivero-Calle I, Sumner E, Fink C, Martinon-Torres F; GENDRES network. Does Viral Co-Infection Influence the Severity of Acute Respiratory Infection in Children? PLoS One. 2016 Apr 20;11(4):e0152481. doi: 10.1371/journal.pone.0152481. eCollection 2016. PMID 27096199
- [Background] Kaforou M, Herberg JA, Wright VJ, Coin LJM, Levin M. Diagnosis of Bacterial Infection Using a 2-Transcript Host RNA Signature in Febrile Infants 60 Days or Younger. JAMA. 2017 Apr 18;317(15):1577-1578. doi: 10.1001/jama.2017.1365. No abstract available. PMID 28418473
- [Background] Wang X, Nijman R, Camuzeaux S, Sands C, Jackson H, Kaforou M, Emonts M, Herberg JA, Maconochie I, Carrol ED, Paulus SC, Zenz W, Van der Flier M, de Groot R, Martinon-Torres F, Schlapbach LJ, Pollard AJ, Fink C, Kuijpers TT, Anderson S, Lewis MR, Levin M, McClure M; EUCLIDS consortium. Plasma lipid profiles discriminate bacterial from viral infection in febrile children. Sci Rep. 2019 Nov 27;9(1):17714. doi: 10.1038/s41598-019-53721-1. PMID 31776453
- [Result] Herberg JA, Kaforou M, Gormley S, Sumner ER, Patel S, Jones KD, Paulus S, Fink C, Martinon-Torres F, Montana G, Wright VJ, Levin M. Transcriptomic profiling in childhood H1N1/09 influenza reveals reduced expression of protein synthesis genes. J Infect Dis. 2013 Nov 15;208(10):1664-8. doi: 10.1093/infdis/jit348. Epub 2013 Jul 29. PMID 23901082
- [Result] Herberg JA, Jones KD, Paulus S, Gormley S, Muir D, Cooper M, Levin M. Comparison of pandemic and seasonal influenza reveals higher mortality and increased prevalence of shock in children with severe h1n1/09 infection. Pediatr Infect Dis J. 2011 May;30(5):438-40. doi: 10.1097/INF.0b013e3182040c90. PMID 21102362
- [Result] Herberg JA, Kaforou M, Wright VJ, Shailes H, Eleftherohorinou H, Hoggart CJ, Cebey-Lopez M, Carter MJ, Janes VA, Gormley S, Shimizu C, Tremoulet AH, Barendregt AM, Salas A, Kanegaye J, Pollard AJ, Faust SN, Patel S, Kuijpers T, Martinon-Torres F, Burns JC, Coin LJ, Levin M; IRIS Consortium. Diagnostic Test Accuracy of a 2-Transcript Host RNA Signature for Discriminating Bacterial vs Viral Infection in Febrile Children. JAMA. 2016 Aug 23-30;316(8):835-45. doi: 10.1001/jama.2016.11236. PMID 27552617
- [Result] Wright VJ, Herberg JA, Kaforou M, Shimizu C, Eleftherohorinou H, Shailes H, Barendregt AM, Menikou S, Gormley S, Berk M, Hoang LT, Tremoulet AH, Kanegaye JT, Coin LJM, Glode MP, Hibberd M, Kuijpers TW, Hoggart CJ, Burns JC, Levin M; Immunopathology of Respiratory, Inflammatory and Infectious Disease Study (IRIS) Consortium and the Pediatric Emergency Medicine Kawasaki Disease Research Group (PEMKDRG). Diagnosis of Kawasaki Disease Using a Minimal Whole-Blood Gene Expression Signature. JAMA Pediatr. 2018 Oct 1;172(10):e182293. doi: 10.1001/jamapediatrics.2018.2293. Epub 2018 Oct 1. PMID 30083721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infection, Inflammation or Allergy | Controls
Started | 818 | 84
Completed | 816 | 84
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infection, Inflammation or Allergy | Controls | Total
Number analyzed (Participants) | 818 | 84 | 902
Age, Customized [Count of Participants; unit: Participants]
  Age at recruitment: <2 years | 467 | 14 | 481
  Age at recruitment: >2 years | 265 | 59 | 324
  Age at recruitment: age not available | 86 | 11 | 97
Sex/Gender, Customized [Count of Participants; unit: Participants]
  gender: male | 318 | 46 | 364
  gender: female | 244 | 29 | 273
  gender: not known | 256 | 9 | 265
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ethnicity: Asian | 63 | 6 | 69
  ethnicity: Black | 85 | 5 | 90
  ethnicity: Mixed race | 32 | 4 | 36
  ethnicity: Other | 30 | 12 | 42
  ethnicity: White | 273 | 24 | 297
  ethnicity: Declined | 71 | 6 | 77
  ethnicity: Ethnicity not available | 264 | 27 | 291
Number of participants with samples taken from sterile site for culture or molecular diagnosis [Count of Participants; unit: Participants] | 818 | 84 | 902

OUTCOME MEASURES:

1. Primary Outcome: What Are the Bacterial and Viral Causes of Acute Illness in Children Presenting to a UK General Hospital, Tertiary Paediatric Infectious Disease Unit and Paediatric Intensive Care Unit?
Description: number of participants with phenotype of definite bacterial or definite viral disease, based on culture or molecular investigations of samples from a sterile site
Time Frame: Participants were monitored for outcome throughout their stay in hospital, and received follow-up review at 10 days
Population: Controls did not present with infectious, inflammatory or allergic conditions - and therefore all patients under the control category had a phenotype of 'healthy' - with none of them meeting criteria for the other phenotype groups (bacterial, viral, inflammatory, uncertain, other).
Measure: Count of Participants; unit: Participants
Arm/Group | Infection, Inflammation or Allergy | Controls
Number analyzed (Participants) | 818 | 84
Participants
  Definite bacterial phenotype | 123 | 0
  Definite viral phenotype | 164 | 0
  Inflammatory phenotype | 41 | 0
  Uncertain phenotype | 450 | 0
  Other phenotype | 40 | 0
  Healthy controls | 0 | 84

ADVERSE EVENTS:
Time Frame: Participants were monitored for all-cause mortality throughout their stay in hospital, and received follow-up review at 10 days if they survived to discharge.
Description: No adverse event data were collected apart from all cause mortality data
Arm/Group | Infection, Inflammation or Allergy | Controls
All-Cause Mortality (participants affected / at risk) | 3/818 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT01022268/Prot_SAP_000.pdf